CLINICAL TRIAL: NCT02793726
Title: The Effects of Large Head Metal on Metal (MOM) Hip Prosthesis on Soft Tissue: Study With 3 Tesla Nuclear Magnetic Resonance (NMR)
Brief Title: The Effects of Large Head MoM Hip Prosthesis on Soft Tissue: Study With 3 Tesla NMR
Acronym: MoM_&_3Tesla
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: MoM and 3 Tesla
Record Dates: First submitted 2016-05-23; First posted 2016-06-08 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2016-06

CONDITIONS: Prostheses and Implants
Keywords: Hip Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Symptomatic: Patients with pain and or other sign of prothesis failure
  Interventions: Procedure: NMR
- Asymptomatic: Patients with regular clinical and radiographic evolution of the implant. No pain
  Interventions: Procedure: NMR

INTERVENTIONS:
Procedure: NMR — NMR

SUMMARY:
Symptomatic and asymptomatic patients wearing Metal on Metal hip prosthesis will be enrolled in the study and periimplant pseudotumors will be searched by means of NMR (Nuclear Magnetic Resonance).

ELIGIBILITY:
Inclusion Criteria:

* Patients wearing MoM hip prosthesis
* Head >= 36 mm

Exclusion Criteria:

* Presence of ferromagnetic implants and/or presence of clinical situations that are not compatible with NMR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients wearing MoM (Metal on Metal) hip prosthesis, head >= 36 mm
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Presence of pseudotumor | at first NMR, between 3 and 6 yrs from surgery
  First NMR will be offered to patients in a period comprised between 3 and 6 yrs from surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli - Laboratorio Tecnologia Medica, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes